CLINICAL TRIAL: NCT00777023
Title: A Phase 3 Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Investigate the Safety and Efficacy of Gabapentin Extended Release (G-ER) Tablets in the Treatment of Vasomotor Symptoms in Postmenopausal Women
Brief Title: Study of Gabapentin Extended Release (G-ER)in the Treatment of Vasomotor (Hot Flashes/Hot Flushes) Symptoms in Postmenopausal Women.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Depomed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: BREEZE 2; 81-0059
Record Dates: First submitted 2008-10-21; First posted 2008-10-22 (Estimated); Results first posted 2012-02-17 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Hot Flashes
Keywords: Hot Flashes; Hot Flushes; Postmenopausal symptoms; Vasomotor symptoms
MeSH Terms: conditions — Hot Flashes | interventions — Gabapentin; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- G-ER 1200 mg (Experimental): Gabapentin extended-release (G-ER) 1200 mg
  Interventions: Drug: Gabapentin Extended-Release (G-ER) 1200 mg
- G-ER 1800 mg (Experimental): Gabapentin extended-release (G-ER) 1800 mg
  Interventions: Drug: Gabapentin Extended-Release (G-ER) 1800 mg
- Sugar Pill (Placebo Comparator): Placebo 1200 mg or 1800 mg
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gabapentin Extended-Release (G-ER) 1200 mg — G-ER 1200 mg daily dosage given as two 600-mg tablets.
  Other Names: Gabapentin
  Arms: G-ER 1200 mg
Drug: Gabapentin Extended-Release (G-ER) 1800 mg — G-ER 1800 mg daily dosage given as one 600-mg tablet in the morning and two 600-mg tablets in the evening.
  Other Names: Gabapentin
  Arms: G-ER 1800 mg
Drug: Placebo — Matching placebo dosages of 1200 mg daily (two 600-mg tablets) and 1800 mg daily (one 600-mg tablet in the morning and two 600-mg tablets in the evening).
  Other Names: Placebo; sugar pill
  Arms: Sugar Pill

SUMMARY:
Depomed's Gabapentin Extended Release is an investigational, extended release formulation of gabapentin that is being studied for the treatment of hot flashes in postmenopausal women

DETAILED DESCRIPTION:
The primary study objective is to assess the efficacy of G-ER dosed in either of the following regimens:

G-ER 1200mg daily (single evening dose)

G-ER 1800mg daily (dosed asymmetrically; 600mg AM/1200mg PM)

compared to placebo in reducing the average daily frequency and severity score of moderate to severe hot flashes in postmenopausal women after 4 weeks and 12 weeks of treatment with a stable dose, compared with the baseline week.

ELIGIBILITY:
Inclusion Criteria:

1. Postmenopausal women aged 18 to 70 years experiencing ≥7 moderate to severe hot flashes per day (or ≥50 per week) accompanied by sweating during previous 30 days or longer.
2. Had amenorrhea for ≥12 months, amenorrhea for 6 to 12 months with serum follicle-stimulating hormone (FSH) levels >40 mIU/mL, or was ≥6 weeks postsurgical bilateral oophorectomy with or without hysterectomy.
3. Willing to discontinue the following: vaginal hormonal products; transdermal or oral estrogen or estrogen/progestin combination; intrauterine progestin; progestin implants; injectable estrogen; topical progesterone cream.
4. Had to have daily average of ≥7 moderate to severe hot flashes and had to complete ≥4 days of diary entries during baseline week to be randomized.
5. If treated with antidepressants, could not have had any changes in drug doses during past month.

Other Inclusions apply.

Exclusion Criteria:

1. Patient treated with a gonadotrophin releasing hormone agonist, anti-estrogens, or aromatase inhibitors within 2 months prior to study entry.
2. Patient treated with estrogen pellets or progestin injectable drugs within 6 months prior to study entry.
3. Patient experience only nighttime hot flashes or worked night shifts on a regular basis.
4. Patient was concurrently treated with gabapentin for other indications. If patient was using gabapentin for treatment of hot flashes, she could be screened after a 7-day washout period provided hot flashes returned.
5. Patient had previously experienced dose-limiting adverse effects that prevented titration of gabapentin to an effective dose.
6. Patient had a hypersensitivity to gabapentin.
7. Patient was in an immunocompromised state.
8. Patient had a malignancy other than basal cell carcinoma within 2 years prior to study entry.
9. Patient had gastric reduction surgery, severe chronic diarrhea, chronic constipation, uncontrolled irritable bowel syndrome, uncontrolled inflammatory bowel disease, or unexplained weight loss.
10. Patient had clinically significant abnormal chemistry or hematology results, or calculated glomerular filtration rate <60 mL/min.
11. Patient had history of substance abuse within year prior to study entry.
12. Patient was concurrently taking morphine.
13. Patient had history of chronic hepatitis B or C, hepatitis within 3 months prior to study entry, or history of human immunodeficiency virus.

Other Exclusions apply.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 565 (Actual)
Dates: Start 2008-10; Primary Completion 2009-07 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (45):
- United States (45):
  - Radiant Research, Birmingham, Alabama
  - Star W Research, Chandler, Arizona
  - Radiant Research, Scottsdale, Arizona
  - May Women's Health Clinic, Little Rock, Arkansas
  - Family Medical Center, Foothill Ranch, California
  - Genesis Center for Clinical Research, San Diego, California
  - San Diego, California
  - Medical Center for Clinical Research, San Diego, California
  - Milestone Medical Research, Inc., Englewood, Colorado
  - Danbury Clinical Research, LLC, Danbury, Connecticut
  - Clinical Research Consulting, LLC, Milford, Connecticut
  - Meridien Research, Bradenton, Florida
  - Meridien Research, Brooksville, Florida
  - Clinical Research of West Florida, Inc., Clearwater, Florida
  - Southeastern Integrated Medical, PL, Gainsville, Florida
  - Sunrise Medical Research, Lauderdale Lakes, Florida
  - University Clinical Research, Inc., Pembroke Pines, Florida
  - Radiant Research - St. Petersburg, Pinellas Park, Florida
  - Atlanta Women's Research Institute, Inc., Atlanta, Georgia
  - Atlanta West Women's Center, Douglasville, Georgia
  - Physician's Research Group, Indianapolis, Indiana
  - West Bank Women's Health, Marrero, Louisiana
  - ActivMed Practices and Research, Haverhill, Massachusetts
  - Women's Health Care Specialists, PC, Paw Paw, Michigan
  - Saginaw Valley Medical Research Group, LLC, Saginaw, Michigan
  - Aspen Medical Group, Saint Paul, Minnesota
  - Clinical Research Center of Nevada, Las Vegas, Nevada
  - Williamsburg Boro Park ObGyn, PC, New York, New York
  - Pinewest Ob-Gyn, Inc., High Point, North Carolina
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - Radiant Research, Inc., Cincinnati, Ohio
  - Rapid Medical Research, Inc., Cleveland, Ohio
  - Columbus Center for Women's Health Research, Columbus, Ohio
  - Clinical Trials of America, Inc., Eugene, Oregon
  - PMG/OB Gyn Health Center, Medford, Oregon
  - The Clinical Trial Center, LLC, Jenkintown, Pennsylvania
  - Upstate Pharmaceutical Research, Greenville, South Carolina
  - Coastal Carolina Research Center, Inc., Mt. Pleasant, South Carolina
  - Alpha Clinical Research, LLC, Clarksville, Tennessee
  - Clinical Research Investigative Services, LLC, Knoxville, Tennessee
  - Mid-South OB-GYN, PLLC, Memphis, Tennessee
  - Renaissance Clinical Research and Hypertension Clinic, Dallas, Texas
  - InVisions Consultants, LLC, San Antonio, Texas
  - Radiant Research, Inc., Salt Lake City, Utah
  - Advanced Clinical Research, West Jordan, Utah

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 565 patients were randomly assigned to treatment: 190 in G-ER 1800 mg group, 192 in G-ER 1200 mg group, and 183 in placebo group. Of these 565 patients, 559 patients (190 in G-ER 1800 mg group, 186 in 1200 mg group, and 183 in placebo group) received study treatment and were included in intent to treat (ITT) and safety populations.
Period: Overall Study
Arm/Group | G-ER 1200 mg | G-ER 1800 mg | Sugar Pill
Started | 186 (192 patients were randomized, but only 186 received study treatment.) | 190 (190 patients were randomized, and 190 received study treatment.) | 183 (183 patients were randomized, and 183 received study treatment.)
Completed | 151 | 149 | 146
Not Completed | 35 | 41 | 37
Not completed — Adverse Event | 15 | 21 | 8
Not completed — Lack of Efficacy | 1 | 0 | 14
Not completed — Protocol Violation | 2 | 1 | 1
Not completed — Lost to Follow-up | 2 | 3 | 3
Not completed — Death | 0 | 1 | 0
Not completed — Withdrawal by Subject | 7 | 7 | 8
Not completed — Missing data | 1 | 1 | 0
Not completed — Reasons not specified | 4 | 4 | 2
Not completed — Last dose date unknown | 3 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | G-ER 1200 mg | G-ER 1800 mg | Sugar Pill | Total
Number analyzed (Participants) | 186 | 190 | 183 | 559
Age Continuous [Mean (Standard Deviation); unit: years] | 53.1 (7.0) | 53.6 (6.1) | 52.9 (6.0) | 53.2 (6.4)
Age, Customized [Number; unit: participants]
  <65 years | 175 | 181 | 177 | 533
  >=65 years | 11 | 9 | 6 | 26
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 186 | 190 | 183 | 559
  Male | 0 | 0 | 0 | 0
Frequency of hot flashes [Mean (Standard Deviation); unit: Hot flashes] — Number of hot flashes in a 24-hour period.
  Hot flashes
    Mild | 1.1 (2.0) | 1.0 (2.0) | 1.7 (2.9) | 1.2 (2.3)
    Moderate | 6.1 (5.8) | 5.4 (4.0) | 6.2 (5.1) | 5.9 (5.0)
    Severe | 6.7 (5.1) | 6.9 (5.5) | 6.6 (4.9) | 6.8 (5.2)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Average Daily Frequency of Moderate or Severe Hot Flashes After 4 Weeks of Treatment
Description: Mean change from baseline in average daily number of moderate or severe hot flashes at stable dose week (SDW) 4 of treatment relative to placebo; last observation carried forward (LOCF) analysis
Time Frame: At baseline and 4 weeks of treatment
Population: Intention to treat population
Measure: Least Squares Mean (95% Confidence Interval); unit: Hot flashes
Arm/Group | G-ER 1200 mg | G-ER 1800 mg | Sugar Pill
Number analyzed (Participants) | 186 | 190 | 183
Hot flashes | -7.0 [-7.77 to -6.19] | -6.9 [-7.68 to -6.08] | -5.4 [-6.18 to -4.46]
Statistical Analysis 1: Comparison: G-ER 1200 mg vs Sugar Pill; Null hypothesis: no treatment differences relative to placebo in mean change from baseline in average daily number of moderate or severe hot flashes at SDW 4; Test type: Superiority or Other; p = 0.0024, ANCOVA — P value for pairwise test of difference of least square mean change from baseline between G-ER 1200 mg and placebo groups based on F test of type III analysis; Mean Difference (Net) = -1.61, 97.5% CI 2-sided [-2.80 to -0.42], Standard Error of Mean 0.53
Statistical Analysis 2: Comparison: G-ER 1800 mg vs Sugar Pill; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0040, ANCOVA — P value for pairwise test of difference of least square mean change from baseline between G-ER 1800 mg and placebo groups based on F test of type III analysis; Mean Difference (Net) = -1.51, 97.5% CI 2-sided [-2.69 to -0.33], Standard Error of Mean 0.52

2. Primary Outcome: Change From Baseline in Average Daily Frequency of Moderate or Severe Hot Flashes After 12 Weeks of Treatment
Description: Mean change from baseline in average daily number of moderate or severe hot flashes at stable dose week (SDW) 12 of treatment relative to placebo; last observation carried forward (LOCF) analysis
Time Frame: At baseline and 12 weeks of treatment
Population: Intent to treat population
Measure: Least Squares Mean (95% Confidence Interval); unit: Hot flashes
Arm/Group | G-ER 1200 mg | G-ER 1800 mg | Sugar Pill
Number analyzed (Participants) | 186 | 190 | 183
Hot flashes | -7.7 [-8.50 to -6.97] | -7.3 [-8.06 to -6.52] | -6.2 [-6.96 to -5.38]
Statistical Analysis 1: Comparison: G-ER 1200 mg vs Sugar Pill; Null hypothesis: no treatment differences relative to placebo in mean change from baseline in average daily number of moderate or severe hot flashes at SDW 12; Test type: Superiority or Other; p = 0.0024, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -1.56, 97.5% CI 2-sided [-2.72 to -0.41], Standard Error of Mean 0.51
Statistical Analysis 2: Comparison: G-ER 1800 mg vs Sugar Pill; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0281, ANCOVA — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Net) = -1.12, 97.5% CI 2-sided [-2.26 to 0.02], Standard Error of Mean 0.51

3. Primary Outcome: Change From Baseline in Average Daily Severity Score of Moderate or Severe Hot Flashes After 4 Weeks of Treatment
Description: Mean change from baseline in average daily severity score of moderate or severe hot flashes at stable dose week (SDW) 4 of treatment relative to placebo; last observation carried forward (LOCF) analysis.
  Severity of hot flashes is scored on a scale of 1 to 3 where 1=mild, 2=moderate, 3=severe.
Time Frame: At baseline and 4 weeks of treatment
Population: Intent to treat population
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | G-ER 1200 mg | G-ER 1800 mg | Sugar Pill
Number analyzed (Participants) | 186 | 190 | 183
Units on a scale | -0.5 [-0.63 to -0.40] | -0.6 [-0.76 to -0.53] | -0.4 [-0.49 to -0.25]
Statistical Analysis 1: Comparison: G-ER 1200 mg vs Sugar Pill; Null hypothesis: no treatment differences relative to placebo in mean change from baseline in average daily severity score of moderate or severe hot flashes at SDW 4; Test type: Superiority or Other; p = 0.0608, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -0.15, 97.5% CI 2-sided [-0.32 to -0.03], Standard Error of Mean 0.08
Statistical Analysis 2: Comparison: G-ER 1800 mg vs Sugar Pill; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0003, ANCOVA — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Net) = -0.28, 97.5% CI 2-sided [-0.45 to -0.11], Standard Error of Mean 0.08

4. Primary Outcome: Change From Baseline in Average Daily Severity Score of Moderate or Severe Hot Flashes After 12 Weeks of Treatment
Description: Mean change from baseline in average daily severity score of moderate or severe hot flashes at stable dose week (SDW) 12 of treatment relative to placebo; last observation carried forward (LOCF) analysis.
  Severity of hot flashes is scored on a scale of 1 to 3 where 1=mild, 2=moderate, 3=severe.
Time Frame: At baseline and 12 weeks of treatment
Population: Intent to treat population
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | G-ER 1200 mg | G-ER 1800 mg | Sugar Pill
Number analyzed (Participants) | 186 | 190 | 183
Units on a scale | -0.8 [-0.90 to -0.61] | -0.8 [-0.97 to -0.68] | -0.5 [-0.69 to -0.39]
Statistical Analysis 1: Comparison: G-ER 1200 mg vs Sugar Pill; Null hypothesis: no treatment differences relative to placebo in mean change from baseline in average daily severity score of moderate or severe hot flashes at SDW 12; Test type: Superiority or Other; p = 0.0280, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -0.21, 97.5% CI 2-sided [-0.43 to 0.00], Standard Error of Mean 0.10
Statistical Analysis 2: Comparison: G-ER 1800 mg vs Sugar Pill; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0026, ANCOVA — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Net) = -0.29, 97.5% CI 2-sided [-0.51 to -0.07], Standard Error of Mean 0.10

ADVERSE EVENTS:
Time Frame: Adverse events collected for total of 13 weeks: from baseline to end of stable dosing week (SDW) 12 (treatment Week 13; end-of-treatment period).
Description: Adverse event collection began at baseline and continued through Week 14 follow-up phone call; serious adverse events followed for 30 days after study completion.
Arm/Group | G-ER 1200 mg | G-ER 1800 mg | Sugar Pill
Serious Adverse Events (participants affected / at risk) | 2/186 | 2/190 | 2/183
Other Adverse Events (participants affected / at risk) | 70/186 | 83/190 | 29/183
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | G-ER 1200 mg (N=186) | G-ER 1800 mg (N=190) | Sugar Pill (N=183)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Overdose; attempted suicide (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Meniscus lesion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | G-ER 1200 mg (N=186) | G-ER 1800 mg (N=190) | Sugar Pill (N=183)
Nausea (Gastrointestinal disorders) | 6 (6) | 14 (14) | 3 (3)
Dizziness (Nervous system disorders) | 32 (32) | 36 (36) | 5 (5)
Headache (Nervous system disorders) | 9 (9) | 14 (14) | 14 (14)
Somnolence (Nervous system disorders) | 13 (13) | 16 (16) | 6 (6)
Sedation (Nervous system disorders) | 10 (10) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI agrees that the sponsor shall have the right to the first publication of the results of the study which is intended to be a joint, multi-center publication. Following the first publication, the PI may publish data or results from the study, provide however PI submits the proposed publication to sponsor for review at least 60 days prior to the date of the proposed publication. Sponsor may remove any information that is considered confidential and/or proprietary other than study data.